CLINICAL TRIAL: NCT04571931
Title: Parental Knowledge, Attitude and Practice Towards Oral Health of Their Children in Relation to Caries Experience
Brief Title: Parental Knowledge, Attitude and Practice Towards Oral Health of Their Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Ibrahim Saeed Eldirdiri, principal investigator, Cairo University
Other Study IDs: oral health questionnaire
Record Dates: First submitted 2020-09-27; First posted 2020-10-01 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the parental knowledge, attitude and practice towards oral health of their children in relation to caries experience.

DETAILED DESCRIPTION:
Primary teeth are important as much as permanent teeth. Dental plaque is considered the major cause of dental diseases, it begins to adhere to the teeth after eruption. Therefore, regular dental care for children becomes essential. Children at preschool age lack the awareness of primary teeth importance, the knowledge in dental health care and the ability to maintain adequate oral health. Hence, it is the parents' responsibility to take care of their children's teeth in collaboration with dentists and their advices.

A good understanding of the parental knowledge, attitudes, beliefs and awareness regarding oral health is essential for the effectiveness of oral health promotion efforts aim at improving the dental health of young children. It has been found that the more positive the attitude of parents is towards dentistry; the better their children's dental health status.

Children from low-income and underprivileged families have been found to have high caries prevalence and poor oral health. Therefore, it is important to assess the knowledge and attitude of parents, as their behaviour towards their children oral health is of a huge impact. This may also have implications on early dental visits aimed for prevention rather than restorative treatment. So, parents' knowledge and attitude have a significant influence on the children's dental and gingival health. Lack of parental knowledge and positive attitudes regarding primary teeth create barriers to early preventive dental care.

In addition, studying and understanding parental dental knowledge and attitude would be of a good help in effective planning for well-targeted dental health promotional campaigns by shedding the light on the knowledge gaps and negative attitudes of the parents regarding dental health

ELIGIBILITY:
Inclusion criteria:

* Parents of children with Primary dentition.

Exclusion criteria:

* Parents of children with psychological problems.
* Parents of children with chronic illness.
* Parents who refuse to participate.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents of preschool children who visiting the outpatient clinic of Pediatric Dentistry and Dental Public Health Department at the Faculty of Dentistry, Cairo University, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Parental knowledge towards oral health | through study completion, an average of one year.
  will be assessed Out of which 10 questions

SECONDARY OUTCOMES:
Parental attitude towards oral health | through study completion, an average of one year.
  will be assessed Out of which 6 questions.
Parental practices towards oral health | through study completion, an average of one year
  will be assessed Out of which 9 questions.
Caries experience of children | through study completion, an average of one year
  using (dmf) caries index.